CLINICAL TRIAL: NCT05400928
Title: The Effect and Safety of Pulsed Field Ablation (PFA) in Patients With Paroxysmal Atrial Fibrillation (PAF)-A Prospective Multicenter Single-arm Study
Brief Title: The Effect and Safety of Pulsed Field Ablation (PFA) in Patients With Paroxysmal Atrial Fibrillation (PAF)
Acronym: ESPFA-CN21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Jiangxi Provincial People's Hopital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Central South University (Other); Second Affiliated Hospital of Nanchang University (Other); Zhongshan Hospital Xiamen University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JJETCT2021002
Record Dates: First submitted 2021-12-01; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Pulsed Field Ablation; Paroxysmal; Ablation; Atrial fibrillation; ring-shaped ablation catheter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-dimensional Directed Pulsed Field Ablation (Experimental): Paroxysmal atrial fibrillation will be ablated with ring-shaped pulsed field ablation catheter directed by integrated three-dimensional mapping system
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — pulmonary vein isolation will be performed with ring-shaped pulsed field ablation catheter directed by integrated three-dimensional mapping system

SUMMARY:
This study is aimed to evaluate the Efficacy and Safety of Pulsed Field Ablation (PFA) in Patients with Paroxysmal Atrial Fibrillation (PAF)

DETAILED DESCRIPTION:
This clinical trial is a prospective, multi-center and single-arm Study. It will be carried out in 3 or more clinical trial institutions, and eligible patients with paroxysmal atrial fibrillation are enrolled. For those patients recruited, pulmonary vein isolation will be performed using pulsed field ablation device (Sichuan Jinjiang Electronic Technology Co., Ltd. Chengdu, China). The safety and efficacy of pulsed field ablation(PFA) in Patients with Paroxysmal Atrial Fibrillation (PAF) will be studied using ring-shaped pulsed field ablation catheter

ELIGIBILITY:
Inclusion Criteria:

Paroxysmal Atrial Fibrillation (PAF)

Exclusion Criteria:

1. A history of atrial fibrillation ablation;
2. Left ventricular ejectfraction(LVEF)<35%
3. Left Atrium(LA)（echocardiography）>55mm
4. Thrombus in the left atrial or heart before surgery
5. New York Heart Association(NYHA) grade Ⅲ-Ⅳ
6. second or third degree atrioventricular block
7. Significant congenital heart defects (e.g. atrial septal defect or severe pulmonary vein stenosis, but except foramen ovale)
8. Prosthetic valves
9. Pacemakers or defibrillators (ICD)
10. Hypertrophic cardiomyopathy, chronic obstructive pulmonary disease or myxoma
11. Symptomatic carotid stenosis
12. Untreated or uncontrolled hyperthyroidism or hypothyroidism
13. Systemic active infection
14. Renal failure with obvious bleeding tendency or undergoing hemodialysis
15. Myocardial infarction or any cardiac intervention/open surgery within 3 months
16. Stroke or transient ischemic attack within 6 months
17. Obvious contraindication for interventional surgery who were determined by the investigator to be unable to undergo ablation
18. Pregnant or lactating women or those who planned to have a family during the study period
19. Have participated in clinical trials of other drugs or medical devices within 3 months
20. Unsuitable to participate in this clinical trial by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Immediate success rate | during procedure
  Procedural success for PAF is defined as the achievement of complete pulmonary venous electrical isolation

SECONDARY OUTCOMES:
Procedural success rate at 12 months after procedure | between 3 months and 12 months after ablation
  Procedural success for PAF was defined as the absence of atrial fibrillation/atrial flutter/atrial tachycardia (duration ≥30s) without antiarrhythmic drugs between 3 months and 12 months after ablation
The occurrence of hospitalizations or emergency department visit due to symptoms of atrial arrhythmia at 6-month and 12-month follow-up | at 6-month and 12-month
  The occurrence of hospitalizations or emergency department visit due to symptoms of atrial arrhythmia at 6-month and 12-month of follow-up
Evaluation of pulsed electric field ablation instrument | baseline
  operational stability; Hardware Connection validity; Software operability; degree of satisfaction
Evaluation of a disposable cardiac pulsed electric field ablation catheter | baseline
  Whether the catheter can reach its desired location smoothly; X ray and shadow;development is clear; Whether the conduit bend is adjustable; Whether the electrophysiological signal is clear and stable; When used together with the mapping system, whether mapping and 3D modeling can be carried out; When used in conjunction with the mapping system, can the catheter be located; Is it possible to stimulate normally; Whether the ablation can be performed normally; Were there any blood clots after withdrawal; Is the tube body intact after withdrawal from the body; Surgeon satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Daowen Wang, PhD, Principal Investigator — Tongji Hospital Wuhan, Hubei China
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansour M, Heist EK, Agarwal R, Bunch TJ, Karst E, Ruskin JN, Mahapatra S. Stroke and Cardiovascular Events After Ablation or Antiarrhythmic Drugs for Treatment of Patients With Atrial Fibrillation. Am J Cardiol. 2018 May 15;121(10):1192-1199. doi: 10.1016/j.amjcard.2018.01.043. Epub 2018 Feb 12. PMID 29571722
- [Background] Hakalahti A, Biancari F, Nielsen JC, Raatikainen MJ. Radiofrequency ablation vs. antiarrhythmic drug therapy as first line treatment of symptomatic atrial fibrillation: systematic review and meta-analysis. Europace. 2015 Mar;17(3):370-8. doi: 10.1093/europace/euu376. Epub 2015 Feb 1. PMID 25643988
- [Background] Reddy VY, Koruth J, Jais P, Petru J, Timko F, Skalsky I, Hebeler R, Labrousse L, Barandon L, Kralovec S, Funosako M, Mannuva BB, Sediva L, Neuzil P. Ablation of Atrial Fibrillation With Pulsed Electric Fields: An Ultra-Rapid, Tissue-Selective Modality for Cardiac Ablation. JACC Clin Electrophysiol. 2018 Aug;4(8):987-995. doi: 10.1016/j.jacep.2018.04.005. Epub 2018 May 11. PMID 30139499
- [Background] Koruth JS, Kuroki K, Iwasawa J, Viswanathan R, Brose R, Buck ED, Donskoy E, Dukkipati SR, Reddy VY. Endocardial ventricular pulsed field ablation: a proof-of-concept preclinical evaluation. Europace. 2020 Mar 1;22(3):434-439. doi: 10.1093/europace/euz341. PMID 31876913
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Maor E, Sugrue A, Witt C, Vaidya VR, DeSimone CV, Asirvatham SJ, Kapa S. Pulsed electric fields for cardiac ablation and beyond: A state-of-the-art review. Heart Rhythm. 2019 Jul;16(7):1112-1120. doi: 10.1016/j.hrthm.2019.01.012. Epub 2019 Jan 11. PMID 30641148
- [Background] Sugrue A, Vaidya V, Witt C, DeSimone CV, Yasin O, Maor E, Killu AM, Kapa S, McLeod CJ, Miklavcic D, Asirvatham SJ. Irreversible electroporation for catheter-based cardiac ablation: a systematic review of the preclinical experience. J Interv Card Electrophysiol. 2019 Sep;55(3):251-265. doi: 10.1007/s10840-019-00574-3. Epub 2019 Jul 3. PMID 31270656
- [Background] Jourda F, Providencia R, Marijon E, Bouzeman A, Hireche H, Khoueiry Z, Cardin C, Combes N, Combes S, Boveda S, Albenque JP. Contact-force guided radiofrequency vs. second-generation balloon cryotherapy for pulmonary vein isolation in patients with paroxysmal atrial fibrillation-a prospective evaluation. Europace. 2015 Feb;17(2):225-31. doi: 10.1093/europace/euu215. Epub 2014 Sep 3. PMID 25186456
- [Background] Iwasawa J, Koruth JS, Petru J, Dujka L, Kralovec S, Mzourkova K, Dukkipati SR, Neuzil P, Reddy VY. Temperature-Controlled Radiofrequency Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Aug 1;70(5):542-553. doi: 10.1016/j.jacc.2017.06.008. PMID 28750697
- [Background] Buist TJ, Adiyaman A, Smit JJJ, Ramdat Misier AR, Elvan A. Arrhythmia-free survival and pulmonary vein reconnection patterns after second-generation cryoballoon and contact-force radiofrequency pulmonary vein isolation. Clin Res Cardiol. 2018 Jun;107(6):498-506. doi: 10.1007/s00392-018-1211-9. Epub 2018 Feb 6. PMID 29411114
- [Background] Furnkranz A, Brugada J, Albenque JP, Tondo C, Bestehorn K, Wegscheider K, Ouyang F, Kuck KH. Rationale and Design of FIRE AND ICE: A multicenter randomized trial comparing efficacy and safety of pulmonary vein isolation using a cryoballoon versus radiofrequency ablation with 3D-reconstruction. J Cardiovasc Electrophysiol. 2014 Dec;25(12):1314-20. doi: 10.1111/jce.12529. Epub 2014 Nov 12. PMID 25146732
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505